CLINICAL TRIAL: NCT03160560
Title: Efficacy of ClōSYS® Oral Rinse Products in Human Subjects in Controlling Oral Malodor
Brief Title: Controlling Oral Malodor by ClōSYS® Oral Rinse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rowpar Pharmaceuticals, Inc. (Industry)
Collaborators: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LLUSD-RPR-Malodor-ADA-2016
Record Dates: First submitted 2017-05-10; First posted 2017-05-19 (Actual); Results first posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Oral Malodor
MeSH Terms: interventions — Mouthwashes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Test-Unflavored Rinse (Active Comparator): CloSYS Oral Rinse product containing 0.1% stabilized chlorine dioxide (sodium chlorite) in aqueous solution.
  Interventions: Drug: ClōSYS® Unflavored Rinse
- Test-Flavored Rinse (Active Comparator): CloSYS Oral Rinse product containing 0.1% stabilized chlorine dioxide (sodium chlorite) in aqueous solution with mint flavoring.
  Interventions: Drug: ClōSYS® Flavored Rinse
- Placebo (Placebo Comparator): CloSYS Oral Rinse product (no chlorine dioxide)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ClōSYS® Unflavored Rinse — Subjects in Test group will receive ClōSYS® Unflavored Rinse.
  Other Names: Mouth rinse
  Arms: Test-Unflavored Rinse
Drug: ClōSYS® Flavored Rinse — Subjects in Test group will receive ClōSYS® Flavored Rinse.
  Other Names: Mouth rinse
  Arms: Test-Flavored Rinse
Other: Placebo — Subjects in Placebo group will receive Placebo Rinse.
  Arms: Placebo

SUMMARY:
The purpose of this Study is to assess the efficacy of two ClōSYS Oral Rinse products in human subjects in controlling oral malodor in partial fulfillment of the requirements for American Dental Association's (ADA) requirement for obtaining ADA Seal for malodor.

DETAILED DESCRIPTION:
Study Design:

The products used in the study are: ClōSYS Alcohol-Free Oral Rinse (also referred as ClōSYS Unflavored Oral Rinse) and ClōSYS justRIGHT MILD MINT Oral Rinse (also referred as ClōSYS Flavored Oral Rinse or Gentle Mint Flavored Oral Rinse). This is an in-vivo, eight-week, a single-center, randomized, double-blind (subject/investigator), 2-way cross-over design clinical study. There are two independent groups. Each subject of each group gets crossed over to the other sub-group within a same group after the washout period. Each group has their own control group. In the first phase, 25 subjects (50%) of each group are randomly assigned to the active group; the other 25 subjects are assigned to the control group. In the second phase, the participants will be crossed over within sub-group assignment. The Study enrolled 100 subjects, aged 21 to 65 years, with a slight to strong intrinsic oral malodor, as determined by a panel of trained odor judges calibrated and standardized using a range of standard odorants sufficient to reflect the different patterns of nose receptors.

Study Plan:

Subjects will receive verbal and written oral hygiene instructions, and either one bottle (16 oz. each) of ClōSYS Unflavored Oral Rinse, ClōSYS Flavored Oral Rinse- or Placebo Oral Rinse each week. Subjects will also receive measuring cups for dispensing the rinse and a diary log for recording usage (the Oral Hygiene Kit) for use during the treatment. After a 2-week wash out period, each subject will receive another bottle of oral rinse according to their group assignment.

Subjects will be instructed to rinse twice a day, each in the morning and in the evening, with 15 mL mouth rinse for 30 seconds. They will note in their patient's log the date and time of rinsing.

Subjects will be instructed to continue with their normal oral hygiene practices, including tooth brushing but omitting any use of oral rinses or mouthwashes except for the Study materials. The subjects also will be instructed not to use other non-study related products such as breath mints, lozenge, gums, etc. as well as refraining from elective dental procedures during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the Informed Consent.
* Must be able to follow verbal/written instructions.
* Between 21 to 65 years of age, male or female.
* Has normal oral interior cheek wall tissues.
* In good general health.
* Should not have any severe or debilitating disease that may impede participation.
* Average organoleptic intensity rating of at >2.6 but <4.5 on an intensity scale of 0-5.

Exclusion Criteria:

* Pregnant or nursing.
* Diagnosis of Xerostomia, including medication induced Xerostomia.
* Oral or extraoral piercing that interferes with the clinical assessments in the mouth.
* Fixed or removable oral appliance.
* Advanced periodontal disease or excessive gingival recession.
* Known allergy or sensitivity to study products.
* Unwilling to abstain from all oral hygiene products other than those prescribed for the study.
* Heavy deposits of calculus, either supragingival and/or subgingival.
* History of severe transmittable infectious disease e.g. hepatitis, HIV, tuberculosis.
* Medical or dental condition that would be unduly affected by participation in this study.
* Any other condition that may interfere with the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Li, DDS MSD PhD, Principal Investigator — Center for Dental Research, Loma Linda University School of Dentistry

IPD SHARING:
Plan to Share IPD: Yes
Results are available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: unlimited
Access Criteria: Request

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study panelists were recruited by placing IRB-approved advertisements in the the Loma Linda University newsletter and local communities. Potential subjects were interviewed by telephone and screened for their eligibility to participate in the study.
Groups:
- Test-Unflavored Rinse, Then Placebo: Participants received ClōSYS® Unflavored Rinse for use for 3 weeks. After a 2-week washout period, the subjects received Placebo rinse for use for 3 weeks.
- Test-Flavored Rinse, Then Placebo: Participants received ClōSYS® Flavored Rinse for use for 3 weeks. After a 2-week washout period, the subjects received Placebo rinse for use for 3 weeks.
- Placebo, Then Flavored Rinse: Participants received Placebo for use for 3 weeks. After a 2-week washout period, the subjects received ClōSYS® Flavored Rinse rinse for use for 3 weeks.
- Placebo, Then Unflavored Rinse: Participants received Placebo for use for 3 weeks. After a 2-week washout period, the subjects received ClōSYS® Unflavored Rinse rinse for use for 3 weeks.
Period: First Intervention (3 Weeks)
Arm/Group | Test-Unflavored Rinse, Then Placebo | Test-Flavored Rinse, Then Placebo | Placebo, Then Flavored Rinse | Placebo, Then Unflavored Rinse
Started | 25 | 25 | 25 | 25
Completed | 23 | 24 | 24 | 25
Not Completed | 2 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0
Period: Washout (2 Weeks)
Arm/Group | Test-Unflavored Rinse, Then Placebo | Test-Flavored Rinse, Then Placebo | Placebo, Then Flavored Rinse | Placebo, Then Unflavored Rinse
Started | 23 | 24 | 24 | 25
Completed | 23 | 24 | 24 | 25
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention (3 Weeks)
Arm/Group | Test-Unflavored Rinse, Then Placebo | Test-Flavored Rinse, Then Placebo | Placebo, Then Flavored Rinse | Placebo, Then Unflavored Rinse
Started | 23 | 24 | 24 | 25
Completed | 22 | 24 | 24 | 25
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Test-Unflavored Rinse, Then Placebo: Participants received ClōSYS® Unflavored Rinse, Then Placebo Unflavored Rinse
- Test-Flavored Rinse, Then Placebo: Subjects received ClōSYS® Flavored Rinse, Then Placebo Flavored Rinse.
- Placebo, Then Flavored Rinse: Subjects in Placebo group received Placebo Rinse, then ClōSYS® Flavored Rinse
- Placebo, Then Unflavored Rinse: Subjects in Placebo group received Placebo Rinse, then ClōSYS® Unflavored Rinse.
- Total: Total of all reporting groups
Arm/Group | Test-Unflavored Rinse, Then Placebo | Test-Flavored Rinse, Then Placebo | Placebo, Then Flavored Rinse | Placebo, Then Unflavored Rinse | Total
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 25 | 25 | 100
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Participant-level, continuous data were collected for participants who did not discontinue the study.
  years
    number analyzed (Participants) | 23 | 24 | 24 | 25 | 96
    (all) | 45.6 (13.5) | 40.6 (13.3) | 38.2 (13.3) | 45.7 (13.9) | 42.5 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex data were only collected from participants that did not elect to discontinue the study.
  Participants
    number analyzed (Participants) | 23 | 24 | 24 | 25 | 96
    Female | 10 | 18 | 16 | 8 | 52
    Male | 13 | 6 | 8 | 17 | 44
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 25 | 25 | 100

OUTCOME MEASURES:

1. Primary Outcome: Change in Malodor as Measured by Organoleptic Score
Description: A 6-level organoleptic score from 0 - 5 will be used. Score of 0 indicating malodor cannot be detected and score of 5 indicating very strong malodor. Breath scores were compared to baseline with malodor intensity reduction recorded as negative.
Time Frame: At baseline and weekly for 3 weeks for each condition and cross-over
Population: All participants
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Unflavored Rinse, Then Placebo: CloSYS Oral Rinse product containing 0.1% stabilized chlorine dioxide (sodium chlorite) in aqueous solution.
  ClōSYS® Unflavored Rinse: Subjects in Test group will receive ClōSYS® Unflavored Rinse, then Placebo.
- Flavored Rinse, Then Placebo: CloSYS Oral Rinse product containing 0.1% stabilized chlorine dioxide (sodium chlorite) in aqueous solution with mint flavoring.
  ClōSYS® Flavored Rinse: Subjects in Test group will receive ClōSYS® Flavored Rinse, then Placebo
- Placebo Flavored, Then Flavored Rinse: CloSYS Oral Rinse product (no chlorine dioxide)
  Placebo: Subjects in Placebo group will receive Placebo Rinse, then Flavored CloSYS Oral Rinse.
- Placebo Unflavored, Then Unflavored Rinse: CloSYS Oral Rinse product containing 0.1% stabilized chlorine dioxide (sodium chlorite) in aqueous solution.
  ClōSYS® Unflavored Rinse: Subjects in Test group will receive Placebo, then ClōSYS® Unflavored Rinse.
Arm/Group | Unflavored Rinse, Then Placebo | Flavored Rinse, Then Placebo | Placebo Flavored, Then Flavored Rinse | Placebo Unflavored, Then Unflavored Rinse
Number analyzed (Participants) | 23 | 24 | 24 | 25
score on a scale
  Baseline | 3.09 (.34) | 3.08 (.38) | 3.03 (.19) | 3.23 (.41)
  Week 1 | 2.90 (.52) | 2.92 (.31) | 3.11 (.46) | 3.19 (.50)
  Week 2 | 2.64 (.48) | 2.78 (.40) | 3.07 (.53) | 3.12 (.43)
  Week 3 | 2.58 (.43) | 2.68 (.51) | 3.07 (.44) | 3.19 (.43)
  Baseline 2-Crossover | 3.44 (.50) | 3.20 (.44) | 3.15 (.42) | 3.14 (.46)
  Week 6: number analyzed (Participants) | 22 | 24 | 24 | 25
  Week 6 | 3.18 (.61) | 3.04 (.49) | 3.17 (.46) | 3.0 (.41)
  Week 7: number analyzed (Participants) | 22 | 24 | 24 | 25
  Week 7 | 3.01 (.59) | 2.94 (.48) | 3.13 (.40) | 3.10 (.5)
  Week 8: number analyzed (Participants) | 22 | 24 | 24 | 25
  Week 8 | 2.96 (.49) | 2.83 (.44) | 3.10 (.40) | 3.09 (.43)
Statistical Analysis 1: Comparison: Flavored Rinse, Then Placebo; Baseline, Week 1, Week 2, Week 3; Test type: Superiority; p < 0.010, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo Flavored, Then Flavored Rinse; Baseline, Week 1, Week 2, Week 3; Test type: Superiority; p = .932, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo Flavored, Then Flavored Rinse; Baseline 2, Week 6, Week 7, Week 8; Test type: Superiority; p = .853, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Flavored Rinse, Then Placebo; Baseline-2, Week 6, Week 7, Week 8; Test type: Superiority; p = .032, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Unflavored Rinse, Then Placebo; Baseline, Week 1, Week 2, Week 3; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo Unflavored, Then Unflavored Rinse; Baseline, Week 1, Week 2, Week 3; Test type: Superiority; p = .750, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Placebo Unflavored, Then Unflavored Rinse; Baseline 2, Week 6, Week 7, Week 8; Test type: Superiority; p = .810, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Unflavored Rinse, Then Placebo; Baseline 2, Week 6, Week 7, Week 8; Test type: Superiority; p = .006, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Eight weeks (the entire course of the study)
Groups:
- Placebo Flavored Rinse; Placebo Unflavored Rinse: Placebo: Subjects in Placebo group will receive Placebo Rinse.
Arm/Group | Test-Unflavored Rinse | Test-Flavored Rinse | Placebo Flavored Rinse | Placebo Unflavored Rinse
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Statistical Analysis Plan (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT03160560/SAP_000.pdf